CLINICAL TRIAL: NCT05402280
Title: Sleep Disturbances in Hospitalized Patients as a Risk Factor for Delirium
Brief Title: Sleep Disturbances and Delirium
Acronym: SLEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ostrava (Other)
Collaborators: University Hospital Ostrava (Other); General University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SLEEP
Record Dates: First submitted 2022-05-19; First posted 2022-06-02 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Sleep Disturbance
Keywords: sleep disruptions; delirium; inpatient; sleep protocol; actigraphy; interventions
MeSH Terms: conditions — Parasomnias; Delirium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Qualitative study (No Intervention): 15 nurses (direct care nurses, nurse managers) and 5 patients, to investigate experiences and compare attitudes and opinions concerning the need for and quality of sleep in hospitalized patients.
- Prospective quantitative study (No Intervention): diagnosing predisposition to sleep disturbances: 400 inpatients staying in gene-ral wards: Patients will undergo a serial of structured and standardized questi-onnaires during scheduled: FIRST: on the day of admission and RCSQ during their hospital stay (record length of up to 7 days).
- Retrospective quantitative study (No Intervention): subjective assessment of factors affecting sleep: 600 hospitalized patients (360 patients in general wards, 240 patients in intensive care wards). On the day of discharge, patients will retrospectively assess disruptive factors that could in-fluence the quality of their sleep during their hospital stay by standardized que-stionnaire.
- Interventional study (Other): (subjective and objective assessment of sleep, quality of sleep with respect to delirium, baseline - routine care: PRE phase) implementation of sleep protocol and assess effectiveness (POST phase: determining the effectiveness of imple-mented sleep measures): overal: 2240 patients (1480 general ward, 760 inten-sive care wards.
  Interventions: Behavioral: Sleep protocol

INTERVENTIONS:
Behavioral: Sleep protocol — To investigate the effect of a multicomponent sleep protocol on the quality of sleep hospitalized patients assessed both subjectively and objectively.
  Other Names: Sleep promotion protocol
  Arms: Interventional study

SUMMARY:
Delirium is a frequent and serious problem in hospitalized patients; it is associated with multiple hospital-acquired complications. There is evidence that the incidence of deliri-um may be minimized by multimodal interventions (pain management, shortening the duration of mechanical ventilation, light sedation, avoiding benzodiazepines, routine delirium monitoring, and early mobilization). Even though a clear association between sleep and delirium has not been established, many studies suggest that sleep disturban-ces may be a key risk factor for the development of delirium. Therefore, sleep promoti-on is becoming an integral part of clinical care. The project support the hypothesis that non-pharmacological preventive interventions promoting sleep (sleep protocol) positive-ly influence the quality of sleep and reduce the incidence of delirium in hospitalized patients. This will be verified by qualitative and quantitative research methods, with the quantitative study being divided into three prospective cross-sectional studies and one interventional study. Data will be obtained from 3240 hospitalized patients by combi-ning subjective methods (questionnaire surveys) and objective measurements (acti-graphy). The project outcomes will allow better understanding of the relationship betwe-en sleep and delirium. A set of non-pharmacological preventive interventions promoting sleep will be developed, with a subsidiary aim to potentially reduce the incidence of delirium in hospitalized patients.

DETAILED DESCRIPTION:
Sleep is one of the most important physiological needs. Sleep disturbances have detri-mental effects on practically all systems and may thus prolong recovery of patients. Studies have documented many similarities between clinical and physiological profiles of patients with delirium and sleep disturbances (ischemia/inflammation, hypoxia, neu-rotransmitter imbalance and tryptophan/melatonin metabolism abnormalities). There is still a lack of strong evidence to support the link between poor sleep and delirium, par-ticularly in hospitalized patients, even though available studies suggest that sleep dis-turbances may be a potential key risk factor for its development, which may have a significant clinical impact. Low awareness of the negative impact of sleep disturbances on the organism and the options for improving sleep may influence the attitude of health professionals to fulfilling this basic human need.The aim of the study is to assess the quality of sleep in patients staying in general wards and intensive care units, identify disruptive factors responsible for its reduced quality, evaluate the relationship between sleep quality and delirium and verify the effectiveness of preventive measures (sleep protocol) in clinical practice. The aims of the study will be met by combining the fol-lowing methods qualitative research, a cross-sectional analytical study and an interven-tional study. The quantitative part of the research will be divided into three consecutive cross-sectional analytical studies. The aim of cross-sectional study I will be to assess the diagnostic properties of the selected instrument (FIRST) for identification of patients predisposed to situational sleep disturbances. This will be immediately followed by cross-sectional study II aimed to identify factors most disrupting sleep of hospitalized patients and, subsequently, by cross-sectional study III subjectively and objectively as-sessing sleep quality and its relationship with delirium, this phase also will be an evalua-tion of routine care (PRE phase), which will be smoothly followed by intervention stud-ies.. The quantitative part is divided into the three cross-sectional studies not only to meet the subgoals and ensure seamless continuity but also because of the patient sam-ple. The patient subgroups are diverse, being specified in detail for each study and se-lected based on the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* a hospital stay longer than 24 hours
* a hospital stay longer than 36 hours
* hospitalized for at least 72 hours, without previous sleep disturbances, without cognitive impairment

Exclusion Criteria:

* Patients with cognitive impairment preventing them from cooperating
* Glasgow Coma Scale score below 12
* terminal disease
* previous and current treatment for sleep disturbances
* neurocognitive dysfunction (dementia)
* sedative administration over the last 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3240 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change quality of sleep during hospitalization (subjectively and objectively) | 25 months
  Assessment of quality of sleep using Richards Campbell Sleep Questionnaire (RCSQ) five-item visual analogue scale was designed as an outcome measure for assessing the perception of sleep in patients. The RCSQ contains 5 items (sleep depth, sleep latency, awakenings, returning to sleep and sleep quality) plus noise as an optional item (evaluated separately). Each item is scored by using a 0-100 visual analogue scale. The total score is calculated as the mean of all items, with 0 and 100 representing the worst and best sleep, respectively. Objectively sleep were assed by actigraphy -the method collects and stores data generated by patient movements.

SECONDARY OUTCOMES:
Change of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) | 25 months
  This is a two-step assessment of delirium. The first step is to assess arousal with the Richmond Agitation and Sedation Scale. The second step is assessment of the presence/absence of delirium using four features; delirium is ruled out when none of them is present.
Change of the Confusion Assessment Method (CAM) | 25 months
  The instrument assesses the presence/absence of delirium using four features; delirium is ruled out when none of them is present.
Change of Ford Insomnia Response to Stress Test: FIRST (self-reported) | 4 months
  The instrument comprises 9 items (scenarios) to identify individuals predisposed to situational sleep disturbances. The FIRST consists of 9 items which are scored on a four point-scale. High scores are indicative of greater vulnerability to sleep disruption. Total FIRST scores range from 9 to 36.
Change of Sleep in the Intensive Care Unit Questionnaire (SICQ) (self-reported) | 3 months
  The most widely used instrument for assessing factors causing sleep disturbances in the ICU. The final version contains 27 items divided into 4 dimensions (sleep quality, daytime sleepiness, disruptive factors produce by the healthcare team and environmental disruptive factors). The ratings use a 1-10 Likert scale.
Change of Questionnaire to ascertain the factors affecting sleep during hospitalization (self-reported) | 3 months
  Scale used for measuring disturbances factors. Questionnaire contains 23 items divided into 4 dimensions (factors - physical, physiological, environmental and psychological). The ratings use a 1-4 Likert scale. The following ranges are used to grade the severity of sleep disturbances: mild sleep disturbances range 0 - 30, moderate disturbances 31 - 60 and severe disturbances 61 - 92.
Analyse information about concerning the need for sleep | up to 1 months
  Semi-structured interviews with inpatiens.
Analyse information about compare attitudes and opinions of nurses providing direct care, nurse managers about sleep and his disturbances | up to 1 months
  Semi-structured interviews with nurses.

CONTACTS AND LOCATIONS:
Overall Officials: Darja Jarosova, Study Director — University of Ostrava
Locations (1):
- University of Ostrava, Ostrava, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alessi CA, Martin JL, Webber AP, Alam T, Littner MR, Harker JO, Josephson KR. More daytime sleeping predicts less functional recovery among older people undergoing inpatient post-acute rehabilitation. Sleep. 2008 Sep;31(9):1291-300. PMID 18788654
- [Background] Altman MT, Knauert MP, Murphy TE, Ahasic AM, Chauhan Z, Pisani MA. Association of intensive care unit delirium with sleep disturbance and functional disability after critical illness: an observational cohort study. Ann Intensive Care. 2018 May 8;8(1):63. doi: 10.1186/s13613-018-0408-4. PMID 29740704
- [Background] Bakken LN, Kim HS, Finset A, Lerdal A. Stroke patients' functions in personal activities of daily living in relation to sleep and socio-demographic and clinical variables in the acute phase after first-time stroke and at six months of follow-up. J Clin Nurs. 2012 Jul;21(13-14):1886-95. doi: 10.1111/j.1365-2702.2011.04014.x. Epub 2012 Apr 4. PMID 22486783
- [Background] Bertisch SM, Pollock BD, Mittleman MA, Buysse DJ, Bazzano LA, Gottlieb DJ, Redline S. Insomnia with objective short sleep duration and risk of incident cardiovascular disease and all-cause mortality: Sleep Heart Health Study. Sleep. 2018 Jun 1;41(6):zsy047. doi: 10.1093/sleep/zsy047. PMID 29522193
- [Background] Bihari S, Doug McEvoy R, Matheson E, Kim S, Woodman RJ, Bersten AD. Factors affecting sleep quality of patients in intensive care unit. J Clin Sleep Med. 2012 Jun 15;8(3):301-7. doi: 10.5664/jcsm.1920. PMID 22701388
- [Background] Boyko Y, Toft P, Ording H, Lauridsen JT, Nikolic M, Jennum P. Atypical sleep in critically ill patients on mechanical ventilation is associated with increased mortality. Sleep Breath. 2019 Mar;23(1):379-388. doi: 10.1007/s11325-018-1718-3. Epub 2018 Sep 13. PMID 30215172
- [Background] Delaney LJ, Currie MJ, Huang HC, Lopez V, Van Haren F. "They can rest at home": an observational study of patients' quality of sleep in an Australian hospital. BMC Health Serv Res. 2018 Jul 5;18(1):524. doi: 10.1186/s12913-018-3201-z. PMID 29976191
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Drake C, Richardson G, Roehrs T, Scofield H, Roth T. Vulnerability to stress-related sleep disturbance and hyperarousal. Sleep. 2004 Mar 15;27(2):285-91. doi: 10.1093/sleep/27.2.285. PMID 15124724
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Flannery AH, Oyler DR, Weinhouse GL. The Impact of Interventions to Improve Sleep on Delirium in the ICU: A Systematic Review and Research Framework. Crit Care Med. 2016 Dec;44(12):2231-2240. doi: 10.1097/CCM.0000000000001952. PMID 27509391
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Patel J, Baldwin J, Bunting P, Laha S. The effect of a multicomponent multidisciplinary bundle of interventions on sleep and delirium in medical and surgical intensive care patients. Anaesthesia. 2014 Jun;69(6):540-9. doi: 10.1111/anae.12638. PMID 24813132
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Smith MT, McCrae CS, Cheung J, Martin JL, Harrod CG, Heald JL, Carden KA. Use of Actigraphy for the Evaluation of Sleep Disorders and Circadian Rhythm Sleep-Wake Disorders: An American Academy of Sleep Medicine Systematic Review, Meta-Analysis, and GRADE Assessment. J Clin Sleep Med. 2018 Jul 15;14(7):1209-1230. doi: 10.5664/jcsm.7228. PMID 29991438
- [Background] Wesselius HM, van den Ende ES, Alsma J, Ter Maaten JC, Schuit SCE, Stassen PM, de Vries OJ, Kaasjager KHAH, Haak HR, van Doormaal FF, Hoogerwerf JJ, Terwee CB, van de Ven PM, Bosch FH, van Someren EJW, Nanayakkara PWB; "Onderzoeks Consortium Acute Geneeskunde" Acute Medicine Research Consortium. Quality and Quantity of Sleep and Factors Associated With Sleep Disturbance in Hospitalized Patients. JAMA Intern Med. 2018 Sep 1;178(9):1201-1208. doi: 10.1001/jamainternmed.2018.2669. PMID 30014139